CLINICAL TRIAL: NCT03587324
Title: Perioperative Risk Factors for the Development of Aspirin Low Response in Patients Undergoing Vascular Surgery.
Brief Title: Perioperative Aspirin Response in Patients Undergoing Vascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Josef Hospital Bochum (Other)
Responsible Party: Principal Investigator, Dr. Thomas Hummel, Thomas Hummel MD, head of the arterial department, vice head of the vascular department, St. Josef Hospital Bochum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Ruhr University of Bochum
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Vascular Surgery Patient With PAD / Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Clopidogrel

ARMS (1):
- Experimental: aspirin, clopidogrel (Experimental): Perioperative measurement of ASA and clopidogrel resistance in patients undergoing vascular treatment
  Interventions: Drug: Whole blood aggregometry before and after vascular treatment (ASA/ Clopidogrel).

INTERVENTIONS:
Drug: Whole blood aggregometry before and after vascular treatment (ASA/ Clopidogrel). — To identify possible risk factors demographic data, concomitant medication, laboratory parameters, co-morbidities, severity of the condition and the type of procedure performed are documented.
  Other Name: ASA (aspirin), Clopidogrel (Plavix)

SUMMARY:
Reduced antiplatelet activity (low response (LR)/high on-treatment platelet reactivity (HPR)) of aspirin (ALR) or clopidogrel (CLR) is associated with an increased risk of thromboembolic events. The prevalence figures for low-responders reported in the literature vary widely and there have been few investigations in vascular surgery patients to date. The aim of this prospective monocentric study was to increase the evidence base on vascular surgery patients and to detect any changes in the response following vascular surgery procedures.

DETAILED DESCRIPTION:
The activity of aspirin (acetylsalicylic acid, ASA) and clopidogrel is measured by whole blood impedance aggregometry using a multiple electrode aggregometer (Multiplate). The agonists used are arachidonic acid for aspirin and adenosine diphosphate (ADP) for clopidogrel. Vascular patients requiring treatment for peripheral artery disease (PAD) and/or carotid stenosis are included in the study. To identify possible risk factors demographic data, concomitant medication, laboratory parameters, co-morbidities, severity of the condition and the type of procedure performed are documented. In addition, a follow-up aggregometry is performed after completion of the vascular procedure.

ELIGIBILITY:
Inclusion Criteria:

• Vascular patients requiring treatment for peripheral artery disease (PAD) and/or carotid stenosis are included in the study.

Exclusion Criteria:

* non-adherence to the antiplatelet medication
* abnormal platelet count in patients,
* current gastrointestinal disorders,
* current infections,
* serious concomitant medical conditions (such as recent gastrointestinal bleeding, cancer, severe cardiac or liver disorders)
* known bleeding or coagulation disorders,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Were Responders or Low-Responders of Antiplatelet Therapy as a Result of Whole Blood Aggregometry Testing | 2 years
  In patients treated with aspirin and clopidogrel aggregometry was performed and depending on the results the patients were either responder or low-responder of antiplatelet therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of vascular surgery, St. Josef Hospital, Ruhr University of Bochum, Bochum, North Rhine-Westphalia, Germany